CLINICAL TRIAL: NCT03171870
Title: Clinical, Radiological Characteristics and Health Related Quality of Life in Idiopathic Pulmonary Fibrosis Patients
Brief Title: Characteristics and Health Related Quality of Life in Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Souad sameh sayed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IPF
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idiopathic Pulmonary Fibrosis (Other): Idiopathic pulmonary fibrosis patients on high resolution computed tomography characterized by presence of reticular opacities often associated with traction bronchiectasis
  Interventions: Diagnostic Test: high resolution computed tomography

INTERVENTIONS:
Diagnostic Test: high resolution computed tomography — high resolution computed tomography is an essential component of the diagnostic pathway in idiopathic pulmonary fibrosis. Unusual interstitial pneumonia is characterized on high resolution computed tomography by the presence of reticular opacities, often associated with traction bronchiectasis

SUMMARY:
Idiopathic pulmonary fibrosis is defined as a specific form of chronic, progressive fibrosing interstitial pneumonia of unknown cause, occurring primarily in older adults, limited to the lungs, and associated with the histopathologic and/or radiologic pattern of usual interstitial pneumonia.

The definition of Idiopathic pulmonary fibrosis requires the exclusion of other forms of interstitial pneumonia including other idiopathic interstitial pneumonias and Interstitial lung disease associated with environmental exposure, medication, or systemic disease.

Prevalence estimates for Idiopathic pulmonary fibrosis have varied from 2 to 29 cases per 100,000 in the general population IPF should be considered in all adult patients with unexplained chronic exertional dyspnea, and commonly presents with cough, bibasilar inspiratory crackles, and finger clubbing.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis should be considered in all adult patients with unexplained chronic exertional dyspnea, and commonly presents with cough, bibasilar inspiratory crackles, and finger clubbing.

High resolution chest computed tomography is an essential component of the diagnostic pathway in Idiopathic pulmonary fibrosis. usual interstitial pneumonia is characterized on high resolution chest computed tomography by the presence of reticular opacities, often associated with traction bronchiectasis.

Patients with interstitial lung disease have poor health-related quality of life. However, whether health-related quality of life differs among different subtypes of interstitial lung disease is unclear.

There is limited research on the health-related quality of life of Idiopathic pulmonary fibrosis patients.

Health-related quality of life deficits should be monitored in clinical practice with Idiopathic pulmonary fibrosis patients and considered when investigating new therapies

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Pulmonary fibrosis will be diagnosed by presence of UIP pattern. Other forms of ILD will be diagnosed using HRCT by presence of Reticular abnormality Honeycombing with or without traction Extensive ground glass abnormality.
* Profuse micronodules.

Exclusion Criteria:

* Patients who refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
To compare Health Related Quality of Life in Idiopathic pulmonary fibrosis patients with other forms of interstitial lung disease | 10 minutes
  St.george respiratory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maha Ghanen, Study Chair — Assiut University; Hoda Makhlouf, Study Chair — Assiut University; Ali Hasan, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han MK, McLaughlin VV, Criner GJ, Martinez FJ. Pulmonary diseases and the heart. Circulation. 2007 Dec 18;116(25):2992-3005. doi: 10.1161/CIRCULATIONAHA.106.685206. PMID 18086941